CLINICAL TRIAL: NCT05557773
Title: The Effects of Core Stabilization Exercises on Balance, Proprioception, and Knee Muscle Strength in Children with Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fuat Gokdemir, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUFGokdemir02
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; core stabilization exercises; balance; proprioception; knee muscle strength

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The control group will be given home based traditional scoliosis exercise training for 8 weeks, 5 days a week for 45 minutes.
  Interventions: Other: Home Based Traditional Scoliosis Exercises
- Training Group (Experimental): In addition to conventional home based traditional scoliosis exercises, patients in this group will also receive core stabilization exercise training for 45 minutes, 5 times in a week for 8 weeks. Every two sessions will be supervised in a clinic per week.
  Interventions: Other: Home Based Traditional Scoliosis Exercises; Other: Core Stability Training

INTERVENTIONS:
Other: Home Based Traditional Scoliosis Exercises — Patients in this group will receive posture exercises, strengthening exercises, diaphragmatic breathing exercises and stretching exercises.
Other: Core Stability Training — Patients in this group will receive traditional scoliosis exercises. In addition, the training group will receive core stabilization exercises for multifidus, diaphragm,erector spines, rectus abdominis, internal and external obliques, quadratus lumborum, iliopsoas, gluteus maximus, and pelvic floor muscles.
  Arms: Training Group

SUMMARY:
Scoliosis can be defined as a 3-dimensional deformity in which the lateral deviation and rotation of the vertebrae occur, as well as changes in the physiological curves of the spine. The gold standard criterion is that the Cobb angle, which determines the lateral deviation of the spine in the frontal plane, is greater than 10°.

Postural control and balance occur as a result of the integration of many sensory information. It is thought that postural control and balance in Adolescent Idiopathic Scoliosis (AIS) patients are adversely affected by biomechanical changes in sensory input, central integration, weight transfer mechanism and the structure of the medulla spinalis. In addition to these, vestibular disorders and proprioceptive losses may have an effect on balance.

Decline in balance reduces the quality of life of individuals with AIS. In addition, exercise has an important place in the treatment of individuals with AIS. In order to get more efficiency from the exercises, it is necessary to improve the balance.

The aim of this study is to evaluate the changes in balance, proprioception, and knee muscle strength of patients, to determine the place of balance exercises in the treatment of individuals with AIS, and to investigate the effect of core stabilization exercises on balance and proprioception in patients with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AIS between the ages of 10-18
* Cobb angle is between 10-40 degrees
* The child's and family's consent to participate in the study
* The child does not receive any other treatment that will affect his scoliosis

Exclusion Criteria:

* Surgical operation in the last 3 months
* Presence of an orthopedic, neurological, systemic disease that will prevent him from exercising
* Having mental, communicative and behavioral disorders that may cause problems understanding commands and questions or performing exercises
* Exercising 3 or more days a week.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Balance | 8 week
  Evaluation of balance with Biodex Balance System
Proprioception | 8 week
  Evaluation of proprioception with Biodex System 3 Pro Multijoint System
Muscle Strength of Knee Flexion / Extension | 8 week
  Muscle Strength of Knee Measurement of isokinetic muscle strength with Biodex System 3Pro Multijoint System Isokinetic Dynamometer.e Flexion / Extension

SECONDARY OUTCOMES:
Balance | 8 week
  Evaluation of balance with Modified Romberg test

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)